CLINICAL TRIAL: NCT02509325
Title: Evaluation of the Parkinson's KinetiGraph Data Logger (PKG) as a Tool to Measure Motor Fluctuations and Support the DBS Eligibility Assessment of Parkinson's Disease Patients.
Brief Title: Parkinson's KinetiGraph as Tool for DBS Eligibility Assessment
Acronym: KITE
Status: Completed | Type: Observational
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Other Study IDs: 1.01.8006
Record Dates: First submitted 2015-07-24; First posted 2015-07-28 (Estimated); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Parkinson's Kinetigraph

SUMMARY:
The purpose of the study is to investigate the feasibility of using the commercially available Parkinson's KinetiGraph Data Logger (PKG) to quantitatively assess motor fluctuations in Parkinson's Disease (PD) patients. A reliable and objective assessment of motor fluctuations would support the general neurologists in the referral of PD patients to the Deep Brain Stimulation (DBS) surgical centers and facilitate the DBS eligibility evaluation of PD patients usually done by the DBS specialists at the DBS surgical centers.

As part of the routine clinical practice, PD patients are referred to the DBS surgical center (clinical site) to optimize their PD treatment and potentially receive a DBS therapy, and the Principal Investigator (PI), a DBS specialist, assesses their DBS eligibility following published expert evaluation criteria and assigns the patient to one of the following two groups (PI assessment):

1. DBS ready, if the patient presents severe motor fluctuations and/or clear dyskinesia history.
2. DBS not-ready, if the patient presents neither severe motor fluctuations, nor clear dyskinesia history.

As part of routine clinical practice, the PKG responsible physician will provide the patient with the PKG to be worn for 6 to 10 days.

Based on the Global Kinetics Corporation (GKC) algorithm applied on the data recorded by the PKG, a GKC representative assigned the patients to one of the above mentioned groups: DBS ready or DBS not-ready.

The primary objective is to evaluate whether the GKC algorithm can differentiate DBS ready from DBS not-ready patients as assessed during the visit at the clinical site by the DBS specialist. The primary endpoint is therefore the percentage of agreement between the PI assessment and the GKC assessment (DBS ready or DBS not-ready) about the DBS eligibility of the PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients are diagnosed with PD.
* Patients are presented to the clinical sites to evaluate DBS candidacy or optimize their PD treatment eventually with DBS therapy.
* Patients are at least 18 years old.
* Patients are able to provide written data release consent as required by Ethics Committee (EC) institutions or local law and regulations.

Exclusion Criteria:

* Patients have restricted movement, e.g. bed bound.
* Patients operate heavy machinery for prolonged periods.
* Patients have serious medical conditions that compromise safety or interfere with mobility in addition to PD (e.g. arthritis and rheumatisms).
* Patients have been already screened by Stimulus or EarlyStimulus questionnaires
* Patients present no response to Levodopa medication or have atypical Parkinsonism.
* Patients have major medical or psychiatric illness other than stable, treated depression or anxiety that may jeopardize the patient's ability to give informed consent, follow study requirements, or that may confound the patient's diagnosis or assessments.
* Patients have major neurological diagnoses other than PD.
* Patients are not capable of following the required clinical instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is represented by Parkinson's Disease (PD) patients who are referred to the DBS surgical center (clinical site) as potential surgical candidate for DBS or to optimize their PD treatment.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Percentage of agreement between the PI assessment and the GKC assessment to differentiate the DBS Ready (DS) from the DBS Not-Ready (DNR) group. | The PI assessment is performed during the examination of the patient by the DBS specialist on the first day of the study. The GKC assessment is calculated once the PKG is returned and it is based on the time period of 6 days of PKG recordings
  The percentage of agreement is the number of patients in the Per Protocol (PP) set for which the GKC assessment is equal to the PI assessment, divided by the total number of patients in the Per Protocol (PP) set and multiplied by 100.

CONTACTS AND LOCATIONS:
Locations (2):
- Centre Hospitalier Universitaire de Grenoble, La Tronche, France
- Universitätsklinikum Würzburg, Würzburg, Germany

REFERENCES:
- [Background] Horne MK, McGregor S, Bergquist F. An objective fluctuation score for Parkinson's disease. PLoS One. 2015 Apr 30;10(4):e0124522. doi: 10.1371/journal.pone.0124522. eCollection 2015. PMID 25928634